CLINICAL TRIAL: NCT05449938
Title: Clinical Evaluation of Impact of Periodontal Phenotype on the Outcome of Scaling and Root Planing in Patients With Periodontitis: A Comparative Interventional Study
Brief Title: Periodontal Phenotype and Scaling and Root Planing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Krishan kant perio
Record Dates: First submitted 2022-06-01; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thick periodontal phenotype (Experimental): Stage II and stage III periodontitis Patient with thick periodontal phenotype will be enrolled using probe transparency method .
  Interventions: Procedure: Scaling and root planing
- Thin periodontal phenotype (Active Comparator): Stage II and stage III periodontitis Patient with thin periodontal phenotype will be enrolled using probe transparency method.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Scaling and root planing involves removal of plaque and calculus on tooth surface.

SUMMARY:
Periodontal phenotype has been recognized as one of the key factors that may potentially impact the outcome of a variety of periodontal surgical and non-surgical procedures. Taking into consideration the inconsistent findings of the studies done in this regard,outcomes of scaling and root planing with respect to periodontal phenotype.

With this aim, the present study would be conducted to assess the influence of periodontal phenotype on outcome of scaling and root planing in periodontitis patients.

DETAILED DESCRIPTION:
AIM: To evaluate the influence of periodontal phenotype on the outcomes of scaling and root planing in periodontitis patients.

OBJECTIVES:

To assess the improvement in pocket probing depth (PPD), clinical attachment level (CAL), bleeding in pocket probing (BOPP), bleeding on marginal probing (BOMP), gingival marginal position (GMP), gingival recession (GR), plaque index (PI), and gingival index (GI) after scaling and root planing (SRP) in periodontitis patients with thin or thick periodontal phenotype.

SETTING: Department of periodontics and oral implantology, PGIDS, Rohtak, Haryana.

STUDY DESIGN: Comparative Interventional study.

TIME FRAME: 12 months (september 2021- August 2022)

POPULATION:

Systemically healthy patients with periodontitis (periodontitis stage II and stage III) and thin/thick periodontal phenotype in maxillary and mandibular incisors will be included.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients with periodontitis (periodontitis stage 2 and stage 3) and thin/thick periodontal phenotype in maxillary and mandibular incisors will be included.

Exclusion Criteria:

* Systemic condition known to affect the course of periodontal disease like diabetes mellitus or immunogenic disorders.
* Patient on anti-inflammatory drugs or antibiotics or history of treatment with medication known to influence periodontal status or healing within last 2 years.
* Current or former smoker or use of tobacco in any form
* History of periodontal treatment in last 2 years
* Crowding in anterior teeth.
* Pregnant or lactating females.
* Individuals with restorations on anterior teeth.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | 6 months
  Change in pocket probing depth from baseline to 6 months
BLEEDING ON POCKET PROBING (BOPP) | 6 months
  Change in bleeding on pocket probing depth from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Krishan Kant, BDS, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES ROHTAK
Locations (1):
- Post Graduate Institute Of Dental Science, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No